CLINICAL TRIAL: NCT00879840
Title: Assessment of Screening Modalities for Gynecologic Cancers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909121; 09-C-N121
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Controls Without Endometrial Cancer; Controls Without Ovarian Cancer
Keywords: Screening; Modalities; Gynecological Cancers
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Females: With endometrial cancer, ovarian cancer, and women undergoing hysterectomy for benign reasons.

SUMMARY:
Background:

* Endometrial and ovarian cancers are, respectively, the fourth and eighth most common cancers among women in the United States. Although some routine Pap tests may detect the presence of cancer cells, there are no convincing early detection approaches for either cancer. Better methods of detection are needed.
* Two possible methods for cancer detection involve samples taken with a tampon or a special kind of brush, called a Tao brush. Researchers would like to know more about how well these methods work.

Objectives:

* To assess the quality of DNA collected by the tampon and Tao brush sampling methods.
* To detect genetic markers in collected DNA and determine if these markers are related to an individual s cancer status.

Eligibility:

* Women age 45 years and older with confirmed or suspected endometrial or ovarian cancer, who will be having surgery.
* A control group of postmenopausal women having surgery for benign gynecological conditions will be included.

Design:

* Shortly before hysterectomy or more extensive procedures to treat either cancer or the benign condition:
* A tampon will be inserted into the vagina to collect cell samples, and removed after 30 minutes.
* After the tampon is removed, the cervix will be swabbed with the Tao brush to collect cell samples.
* Following the hysterectomy, samples of healthy and cancerous tissue will be taken, and tested by researchers.

DETAILED DESCRIPTION:
Background:

Currently, there are no convincing early detection approaches for endometrial and ovarian cancers. Although it is well established that some endometrial and ovarian tumors shed cytologically recognizable cells in routinely prepared Pap tests, it is clear that this approach rarely detects occult tumors. Accordingly, efforts to develop means of collecting biological samples that have high patient acceptability, good sensitivity for detecting early disease, and excellent specificity are needed.

Objectives:

In this project, we want to assess the feasibility of using alternative sampling techniques in combination with molecular assays to detect endometrial and ovarian cancers. We will compare sampling using a Tampon and a sheathed endometrial brush, the Tao brush. We want to assess the quality of DNA extracted from the different samplers. We will assess the correlations between methylation of somatic DNA for a selected marker panel and cancer status.

Eligibility:

We wish to include 117 women age 45 years and older with suspected endometrial cancer, or ovarian cancer, and 53 age-matched (plus/minus 5 years) controls without malignancy, all of whom are referred to surgery at the Mayo clinic.

Design:

We plan to conduct a pilot study of women with confirmed or suspected endometrial cancer, or ovarian cancer, and women treated for benign conditions. DNA will be extracted from samples collected using a vaginal Tampon and an endometrial brushing using an FDA approved device (Tao brush) prior to surgery. A panel of methylation markers will be analyzed from samples yielding sufficient DNA. The results of the methylation analysis will be compared to the final histology for all patients in the study. We will set the detection of methylation at one or more loci in 50% of women in each arm as a technical success.

ELIGIBILITY:
* INCLUSION CRITERIA:
* The study will enroll a total of 170 women consented for hysterectomy. One hundred and seventeen (117) will either have 1) suspected ovarian cancer based on clinical impression, cytologic or histologic diagnoses (effusions, Pap tests or other biopsies), or 2) suspected endometrial cancer based on biopsy diagnoses of atypical endometrial hyperplasia (or its equivalent endometrial intraepithelial neoplasia), endometrial intraepithelial carcinoma (i.e. in-situ/ early serous carcinoma) or carcinoma. Fifty-three (53) will be undergoing definitive treatment for benign conditions (uterine fibroids, benign appearing adnexal pathology and normal CA 125, pelvic floor dysfunction not to exceed grade 1 or 2 uterine descensus). Since the analyzed cancers do not occur in children, they will not be included in this study.

EXCLUSION CRITERIA:

* Surgical candidates for recurrent disease
* Preoperative neoadjuvant chemotherapy or radiotherapy
* History of tubal ligation, salpingitis, or hysterectomy (ovarian cancer patients)
* Control patients who are less than 45 years of age.
* Patients receiving treatment for active endometriosis.
* Cervical stenosis recognized clinically by not accepting the Tao Brush
* Endometrial sampling within 5 days of anticipated surgery
* Prior history of endometrial ablation
* Patients with cervical cancer

Ages: 50 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with endometrial cancer, ovarian cancer, and women undergoing hysterectomy for benign reasons.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2009-04-09 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Endometrial Cancer, ovarian cancer | 1 year
  Histologically confirmed endometrial or ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Mayo Clinic, Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Ries LA. Ovarian cancer. Survival and treatment differences by age. Cancer. 1993 Jan 15;71(2 Suppl):524-9. doi: 10.1002/cncr.2820710206. PMID 8420672
- [Background] Buys SS, Partridge E, Greene MH, Prorok PC, Reding D, Riley TL, Hartge P, Fagerstrom RM, Ragard LR, Chia D, Izmirlian G, Fouad M, Johnson CC, Gohagan JK; PLCO Project Team. Ovarian cancer screening in the Prostate, Lung, Colorectal and Ovarian (PLCO) cancer screening trial: findings from the initial screen of a randomized trial. Am J Obstet Gynecol. 2005 Nov;193(5):1630-9. doi: 10.1016/j.ajog.2005.05.005. PMID 16260202
- [Background] Vine MF, Ness RB, Calingaert B, Schildkraut JM, Berchuck A. Types and duration of symptoms prior to diagnosis of invasive or borderline ovarian tumor. Gynecol Oncol. 2001 Dec;83(3):466-71. doi: 10.1006/gyno.2001.6411. PMID 11733956